CLINICAL TRIAL: NCT06799377
Title: Complications Related to Activity After Both Bone Fractures: Why do we Restrict Activity?
Brief Title: Complications Related To Activity After Pediatric Both Bone Fractures: Exploring the Effects of Activity on Fracture Displacement
Acronym: CRABB-Y
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nathaniel Lempert, Assistant Professor of Pediatric Orthopaedics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 241179
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Forearm Fractures (Both Bone Forearm Fractures, Isolated Ulnar Shaft, Isolated Radial Shaft)

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial with two group that receive different activity restrictions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restricted Activity Group (Active Comparator): This group of patients will be given restricted activity recommendations. They will be told: "Your child has a forearm/wrist fracture. It is unknown if remaining active while in a cast affects the risk of complications after this type of fracture. Your child has been randomized to the "restricted activity" group. We ask that you limit sprinting, jumping, and organized sports during the time of cast immobilization. As a rule of thumb, we recommend "feet on the floor" activities while playing and avoiding playgrounds and gym class if possible. While it is not realistic to restrict a young child entirely, do your best to avoid strenuous or intense exercise until cleared by your physician or nurse practitioner"
  Interventions: Behavioral: Restricted Activity Reccomendations
- Activity (Limited) Group (Active Comparator): This group of patients will be given limited activity recommendations. They will be told "Your child has a forearm/wrist fracture. It is unknown if remaining active while in a cast affects the risk of complications after this type of fracture. Your child has been randomized to the "activity as tolerated" group. Your child may participate in all desired activities except contact sports. Your child does not need to increase his/her activity level but should participate in activities as they feel comfortable doing so. Sprinting, jumping, and organized sports are acceptable as long as your child is not experiencing pain. Your child may use playgrounds and participate in gym class as desired. Do your best to avoid restricting your child from activities unless they are experiencing pain or you have concerns about their safety."
  Interventions: Behavioral: Full Activity/Limited Activity Reccomendations

INTERVENTIONS:
Behavioral: Restricted Activity Reccomendations — Patients in this respective group will be given restricted activity recommendations over the casting period. They will be told "Your child has a forearm/wrist fracture. It is unknown if remaining active while in a cast affects the risk of complications after this type of fracture. Your child has been randomized to the "restricted activity" group. We ask that you limit sprinting, jumping, and organized sports during the time of cast immobilization. As a rule of thumb, we recommend "feet on the floor" activities while playing and avoiding playgrounds and gym class if possible. While it is not realistic to restrict a young child entirely, do your best to avoid strenuous or intense exercise until cleared by your physician or nurse practitioner"
  Arms: Restricted Activity Group
Behavioral: Full Activity/Limited Activity Reccomendations — Patients in this respective group will be allowed to engage in most activities. They will be read "Your child has a forearm/wrist fracture. It is unknown if remaining active while in a cast affects the risk of complications after this type of fracture. Your child has been randomized to the "activity as tolerated" group. Your child may participate in all desired activities except contact sports. Your child does not need to increase his/her activity level but should participate in activities as they feel comfortable doing so. Sprinting, jumping, and organized sports are acceptable as long as your child is not experiencing pain. Your child may use playgrounds and participate in gym class as desired. Do your best to avoid restricting your child from activities unless they are experiencing pain or you have concerns about their safety."
  Arms: Activity (Limited) Group

SUMMARY:
The goal of this randomized clinical study is to understand the effect of activity on the re-displacement of pediatric forearm fractures in patients ages 8-18 years old excluding those with known metabolic bone disease or obvious refracture. The main questions the study aims to answer are:

Does increased activity lead to increased re-displacement rates during the treatment of pediatric forearm fractures? Are there complications associated with increased levels of activity during the treatment of pediatric forearm fractures (skin irritation, need for re-casting, operation)? Do activity restrictions provided for pediatric forearm fractures influence patient activity levels?

Participants will be randomized into activity-restricted vs activity-limited (no contact sports). Some patients will be provided an ActiGraph Activity tracker to monitor patient activity. Every patient will complete a validated activity survey (PAQ) to assess activity at each follow-up appointment. Activity data and any complications will be recorded from time of initial presentation to cast removal.

ELIGIBILITY:
Inclusion Criteria:

* Isolated Distal Radius Metaphyseal Fx (with or without ulna styloid)
* Distal Third (<4 cm from physis) Radius and Ulna fracture (i.e. without obvious physeal involvement)
* Insolated Radial Shaft Fracture (diaphyseal)
* Radial and Ulna Shaft Fracture (diaphyseal)

Exclusion Criteria:

* Initial presentation >7 days from the time of injury
* Pathologic fracture
* Any patient with metabolic bone disease (ex. Osteoporosis, skeletal dysplasias)
* Any patient with known bone fragility condition (ex. Osteogenesis imperfecta)
* If operative treatment is required at initial presentation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Re-Displacement | From Cast Placement to Cast Removal, aproximately 6-8 weeks.
  Re-displacement will be defined as a change in angulation of greater than 10 degrees.

SECONDARY OUTCOMES:
Complications | From casting to cast removal, approximately 6-8 weeks.
  The rate of complications including skin irritation/breakdown, the need for re-casting, and the need for operative management.
Activity Level as measured by patient-completed validated activity surveys (PAQ) | Time of clinic presentation to cast removal, approximately 6-8 weeks.
  Activity levels based on patient-completed validated activity surveys (PAQ)
Activity Level as measured by patient-worn activity trackers | Time of clinic presentation to cast removal, approximately 6-8 weeks
  Activity levels based on patient-worn activity trackers

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Children's Hospital Orthopedics Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not plan to submit to International Committee of Medical Journal Editors (ICMJE)

REFERENCES:
- [Background] Alagoz E, Gulec MA. Factors affecting re-displacement in pediatric forearm fractures and the role of cast indices. Jt Dis Relat Surg. 2020;31(1):95-101. doi: 10.5606/ehc.2020.71523. PMID 32160501
- [Background] Ting BL, Kalish LA, Waters PM, Bae DS. Reducing Cost and Radiation Exposure During the Treatment of Pediatric Greenstick Fractures of the Forearm. J Pediatr Orthop. 2016 Dec;36(8):816-820. doi: 10.1097/BPO.0000000000000560. PMID 26057068
- [Background] Sara Peiffer, Samuel J. Dressler, William L. Hennrikus; Outcomes of Displaced Forearm Fractures in Children Treated With Closed Reduction and Casting and a Loop and Sling Attached to the Cast Proximal to the Fracture Site. Pediatrics March 2021; 147 (3_MeetingAbstract): 798. 10.1542/peds.147.3MA8.798a
- [Background] Sengab A, Krijnen P, Schipper IB. Displaced distal radius fractures in children, cast alone vs additional K-wire fixation: a meta-analysis. Eur J Trauma Emerg Surg. 2019 Dec;45(6):1003-1011. doi: 10.1007/s00068-018-1011-y. Epub 2018 Oct 1. PMID 30276723
- [Background] Knopp BW, Harris M. Pediatric Forearm Fracture Characteristics as Prognostic Indicators of Healing. Cureus. 2023 Feb 7;15(2):e34741. doi: 10.7759/cureus.34741. eCollection 2023 Feb. PMID 36913227

DOCUMENTS (1):
  • Study Protocol (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT06799377/Prot_000.pdf